CLINICAL TRIAL: NCT05486130
Title: PREdiction of CEphalosporinase Producing Enterobacteria During Ventilator-associated Pneumonia for Therapeutic Stewardship
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PRECEPT
Record Dates: First submitted 2022-07-05; First posted 2022-08-03 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ventilator-associated pneumonia is the leading cause of nosocomial infection in the ICU. Cephalosporinase-producing Enterobacteriaceae have an increasing incidence. Infections in cephalosporinase-producing patients require the use of Cefepime during probabilistic antibiotic therapy, the repeated use of which will lead to a significant risk of selection of resistant mutants. The involvement of cephalosporinases being infrequent, the prediction of their presence during a VAP would make it possible to reduce the consumption of Cefepime and thus to take part in the prevention of selection of bacterial mutants resistant to beta-lactams. The main objective of the research is to determine the risk factors for the involvement of cephalosporinase-producing enterobacteria during episodes of ventilator-associated pneumonia (VAP) in hospitalized patients. The secondary objectives are to describe the epidemiology of cephalosporinase-producing enterobacteria in the ICU and to compare the risk factors for the presence of a cephalosporinase-producing germ not without its production being derepressed with those present in situations of cephalosporinase derepression.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years and older
* Patient on mechanical ventilation for more than 48 hours
* Patient with a diagnosis of ventilator-associated lung disease during management according to American Thoracic Society criteria
* French speaking patient

Exclusion Criteria:

* Tracheostomized patient at the time of inclusion
* Limitation of therapies before inclusion in the study
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on mechanical ventilation for more than 48 hours, with a diagnosis of ventilator-associated lung disease during management according to American Thoracic Society criteria.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cephalosporinase-producing enterobacteria during episodes of ventilator-associated pneumonia | 1 month
  This outcome corresponds to the the number of ventilator-associated pneumonias involving cephalosporinase-producing enterobacteria.

SECONDARY OUTCOMES:
Epidemiology of cephalosporinase-carrying enterobacteria in the ICU | 1 month
  This outcome corresponds to the number of pathogens identified in ventilator-associated pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: François PHILIPPART, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Bouadma L, Sonneville R, Garrouste-Orgeas M, Darmon M, Souweine B, Voiriot G, Kallel H, Schwebel C, Goldgran-Toledano D, Dumenil AS, Argaud L, Ruckly S, Jamali S, Planquette B, Adrie C, Lucet JC, Azoulay E, Timsit JF; OUTCOMEREA Study Group. Ventilator-Associated Events: Prevalence, Outcome, and Relationship With Ventilator-Associated Pneumonia. Crit Care Med. 2015 Sep;43(9):1798-806. doi: 10.1097/CCM.0000000000001091. PMID 25978340
- [Background] Wang Y, Eldridge N, Metersky ML, Verzier NR, Meehan TP, Pandolfi MM, Foody JM, Ho SY, Galusha D, Kliman RE, Sonnenfeld N, Krumholz HM, Battles J. National trends in patient safety for four common conditions, 2005-2011. N Engl J Med. 2014 Jan 23;370(4):341-51. doi: 10.1056/NEJMsa1300991. PMID 24450892
- [Background] Damas P, Layios N, Seidel L, Nys M, Melin P, Ledoux D. Severity of ICU-acquired pneumonia according to infectious microorganisms. Intensive Care Med. 2011 Jul;37(7):1128-35. doi: 10.1007/s00134-011-2255-8. Epub 2011 May 26. PMID 21614638
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Crnich CJ, Safdar N, Maki DG. The role of the intensive care unit environment in the pathogenesis and prevention of ventilator-associated pneumonia. Respir Care. 2005 Jun;50(6):813-36; discussion 836-8. PMID 15913471